CLINICAL TRIAL: NCT00610987
Title: Antibiotic Prophylaxis in Orthopaedic Traumatology: A Prospective, Randomized Trial of Duration of Administration
Brief Title: Antibiotic Prophylaxis in Orthopaedic Traumatology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB1089017
Record Dates: First submitted 2008-01-24; First posted 2008-02-08 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Fractures, Closed; Wounds and Injuries
Keywords: Antibiotic Prophylaxis
MeSH Terms: conditions — Fractures, Closed; Wounds and Injuries | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin (Active Comparator): Group I will receive 1-g doses of cefazolin every eight hours for the next 24 hours after surgical repair of the closed limb fracture.
  Interventions: Drug: cefazolin
- Placebo (Placebo Comparator): Group II will receive no additional antibiotic. Instead, they will receive normal saline injection every eight hours as a placebo, after the intraoperative dose(s) of cefazolin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cefazolin — Both groups will receive 1 gram (g) of IV cefazolin prior to incision, per standard protocol at our institution. A 2-g dose of cefazolin will be administered IV for patients weighing more than 80 kg. A second 1-g dose of cefazolin will be given three hours later if the patient is still in the operating room. Upon completion of the surgical procedure, Group I will receive 1-g doses of cefazolin every eight hours for the next 24 hours.
  Other Names: cefazolin brand name = Kefzol
  Arms: Cefazolin
Drug: Placebo — Patients will be randomly assigned to one of two groups. Both groups will receive 1 gram (g) of IV cefazolin prior to incision, per standard protocol at our institution. A 2-g dose of cefazolin will be administered IV for patients weighing more than 80 kg. A second 1-g dose of cefazolin will be given three hours later if the patient is still in the operating room. Upon completion of the surgical procedure, Group II will receive no additional antibiotic. Instead, they will receive normal saline injection every eight hours as a placebo.
  Arms: Placebo

SUMMARY:
It has been established that providing antibiotic prophylaxis after closed fracture fixation with implants or prosthetic devices has beneficial effects. However, the optimal duration of antibiotic prophylaxis after orthopaedic trauma surgery is not well-defined. Most studies comparing single-dose prophylaxis with multiple-dose prophylaxis have not shown beneficial effects of additional doses. Our proposed study is intended to further define the appropriate duration of antibiotic (cefazolin) administration for surgical prophylaxis in the treatment of closed fractures. We will randomly assigned patients into two groups, hopefully differentiated only by the duration of antibiotic administration (single dose vs. 24 hours). We will follow these patients until fracture healing and determine if there is a difference in the incidence of infection.

DETAILED DESCRIPTION:
The proposed study is a prospective, randomized, double-blinded clinical trial intended to further define the appropriate duration of antibiotic (cefazolin) administration for surgical prophylaxis in the internal fixation of closed fractures. Our hypothesis is that there will be no difference in the incidence of infection between single-dose versus 24 hours of antibiotic prophylaxis. The null hypothesis is that multiple-dose antibiotic prophylaxis will have a decreased incidence of infection.

Research Design:

A prospective, randomized, double-blinded clinical trial will be conducted to evaluate the duration of antibiotic prophylaxis. After investigators obtain Institutional Review Board approval, recruited patients will be randomly assigned to one of two groups. Both groups will receive 1 gram (g) of IV cefazolin prior to incision, per standard protocol at our institution. If a tourniquet is used, the cefazolin will be administered at least 10 minutes prior to inflation. A 2-g dose of cefazolin will be administered IV for patients weighing more than 80 kg. A second 1-g dose of cefazolin will be given three hours later if the patient is still in the operating room. Upon completion of the surgical procedure, Group I will receive 1-g doses of cefazolin every eight hours for the next 24 hours. Group II will receive no additional antibiotic. Instead, they will receive normal saline injection every eight hours as a placebo. Group assignments will not be disclosed to the evaluators responsible for clinical examination or to the patients until the end of the study.

Either an orthopaedic surgeon or nurse practitioner will evaluate the patients for the development of a wound infection. Follow-up will occur at 10-14 days, six weeks, 12 weeks, and every six to eight weeks thereafter until bony union occurs. Wound infection will be defined as one or more of the classic signs and symptoms of inflammation (rubor, calor, tumor, dolor) together with purulent drainage at the operative site. Wound infections will be classified either as superficial (infection of the skin or subcutaneous tissue, not communicating with the bone) or deep (infection that reached bone or material implanted for osteosynthesis). Bacteriological cultures will be obtained in the event of infectious complications, but wound infections will be diagnosed clinically.

Several studies have demonstrated that there are numerous patient-related and treatment-related factors that predispose to infectious complications. We will use several of these factors to assign a risk score to each of the enrolled patients. Each factor will be worth one point for a total score ranging from 0 (lowest risk) to 7 (highest risk). The risk factors are: 1) smoking; 2) age >65; 3) diabetes mellitus; 4) obesity (BMI >35); 5) duration of surgery >3 hours; 6) urinary catheterization (0=no catheter, 1=catheter <48 hours, 2=catheter >48 hours).

Statistical evaluation will be conducted by Student's t-test for patient characteristics and chi square analysis for infection rates. The relation between wound infection and the various possible risk factors will be assessed by forward stepwise logistic regression analysis. Significance will be defined at the P < 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older;
* Scheduled for primary osteosynthesis or placement of a prosthetic device in the treatment of closed limb fractures;
* Ability to give informed consent.

Exclusion Criteria:

* Known hypersensitivity to cephalosporins;
* Antimicrobial use or symptoms of infection in the week before surgery;
* Pregnancy;
* Immunosuppressive treatment;
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After IRB approval, patients undergoing ORIF of closed fractures that had a planned postoperative stay of at least 23 hours were randomized to either receiving 23 hours of cefazolin or a placebo.
Pre-assignment Details: After IRB approval, patients undergoing ORIF of closed fractures that had a planned postoperative stay of at least 23 hours were randomized to either receiving 23 hours of cefazolin or a placebo.
Period: Overall Study
Arm/Group | Cefazolin | Placebo
Started | 75 | 71
Completed | 75 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefazolin | Placebo | Total
Number analyzed (Participants) | 75 | 71 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 37 | 92
  >=65 years | 20 | 34 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (19.1) | 50.5 (20.5) | 49.8 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 39 | 69
  Male | 45 | 32 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Wound Infections
Description: The primary endpoint was infection.
Time Frame: at 10-14 days, six weeks, 12 weeks, and every six to eight weeks thereafter until bony union occurs.
Measure: Number; unit: participants
Arm/Group | Cefazolin | Placebo
Number analyzed (Participants) | 75 | 71
participants | 4 | 9
Statistical Analysis 1: Comparison: Cefazolin vs Placebo; Test type: Superiority or Other; p = 0.12, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Cefazolin | Placebo
Serious Adverse Events (participants affected / at risk) | 18/75 | 22/71
Other Adverse Events (participants affected / at risk) | 0/75 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cefazolin (N=75) | Placebo (N=71)
Infections (Infections and infestations) | 15 (15) | 5 (5)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 3 (3)
trauma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
implant problems (Surgical and medical procedures) | 1 (1) | 2 (2)
vascular (Vascular disorders) | 0 (0) | 2 (2)
General disorders including death (General disorders) | 1 (1) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No